CLINICAL TRIAL: NCT01052259
Title: Pilot Study of Cycling Treatment of Deoxyspergualin in Biopsy-proven Chronic Rejection of Kidney Transplantation
Brief Title: Efficacy and Safety of Deoxyspergualin in Renal Transplant Patient With Chronic Rejection
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insufficient patient enrollment
Sponsor: Nippon Kayaku Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SPCR2009
Record Dates: First submitted 2010-01-14; First posted 2010-01-20 (Estimated); Last update posted 2014-01-08 (Estimated); Status verified 2014-01

CONDITIONS: Chronic Rejection
Keywords: Chronic rejection; Kidney; Transplantation; Immunosuppressive
MeSH Terms: interventions — gusperimus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Deoxyspergualin, Treatment, (Experimental)
  Interventions: Drug: Deoxyspergualin

INTERVENTIONS:
Drug: Deoxyspergualin — 100mg/vial as active substance; Deoxyspergualin at 3-5 mg/kg/day by 1-3 iv infusion will be given once a day for 5 to 7 days each cycle every month; Total cycle treatment will be 6.
  Other Names: Spanidin, gusperimus hydrochloride

SUMMARY:
The purpose of this study to examine the efficacy and safety of cycling treatment of deoxyspergualin in renal transplant patients with biopsy-proven chronic rejection.

DETAILED DESCRIPTION:
The primary aim of this study is to investigate the efficacy of deoxyspergualin after the completion of 6 cycles treatment. The efficacy valuables are histological findings in renal grafts, renal function, proteinuria, graft survival, anti-HLA antibody. The safety data are also evaluated in the study.

ELIGIBILITY:
Inclusion Criteria:

* Chronic rejection defined by Banff 2007 criteria

Exclusion Criteria:

* Patients who have recurrent renal diseases and virus-associated renal diseases
* Patients who have initial WBC < 4,000, neutrophil < 1,000 , platelet < 50,000 or Hb < 8g
* Patients who have acute or chronic infection

Ages: 11 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2009-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Histopathological findings by Banff criteria | 6 month after treatment initiation

SECONDARY OUTCOMES:
Renal function, proteinuria, graft survival, anti-HLA antibody, adverse events, serious adverse events (SAE) | 6 and 12 months after treatment initiation

CONTACTS AND LOCATIONS:
Overall Officials: Hiroshi Harada, Chief, Principal Investigator — Sapporo City General Hospital
Locations (8):
- Japan (8):
  - Akita University School of Medicine, Akita, Akita
  - Graduate School of Medicine Sciences, Kyushu University, Fukuoka, Fukuoka
  - Gifu University Graduate School of Medicine, Gifu, Gifu
  - Sapporo City General Hospital, Sapporo, Hokkaido
  - Osaka University Graduate School of Medicine, Suita, Osaka
  - Toda Central General Hospital, Toda, Saitama
  - Toho University Graduate School of Medicine, Ōta-ku, Tokyo
  - Tokyo Women's Medical University, Shinjuku-ku, Tokyo